CLINICAL TRIAL: NCT01266122
Title: Addressing Psychosocial Needs and HIV Risk in Indian MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Tuberculosis Research Centre, India (Other Government); Fenway Community Health (Other)
Responsible Party: Principal Investigator, Steven A. Safren, Director, Behavioral Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R21MH085314-02 (NIH); 5R21MH085314-02 (NIH)
Record Dates: First submitted 2010-11-24; First posted 2010-12-24 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: HIV/STI Risk; HIV/STI Incidence
Keywords: HIV; Psychosocial problems; MSM; India
MeSH Terms: interventions — Behavior Therapy; Psychosocial Intervention; dimethyl sulfone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV/STI voluntary counseling and testing (No Intervention): Participants enrolled in the control arm will receive study assessments only.
- Behavioral intervention (Experimental): Participants enrolled in the experimental condition will receive 4 group sessions and 4 individual sessions over 3 months. This intervention focuses on psychosocial concerns and HIV risk for MSM in India.
  Interventions: Behavioral: Behavioral intervention

INTERVENTIONS:
Behavioral: Behavioral intervention — The behavioral intervention will consist of 4 group sessions and 4 individual sessions over 3 months. The overall focus is on psychosocial concerns and HIV risk.
  Other Names: Psychosocial intervention for MSM in India
  Arms: Behavioral intervention

SUMMARY:
This study will develop and pilot test a combined individual and group-level behavioral HIV prevention intervention for men who have sex with men (MSM) in Chennai, India, addressing HIV risk within the context of broader psychosocial issues, including self-acceptance, substance use and social support.

DETAILED DESCRIPTION:
MSM in India are at increased risk for HIV in a stigmatizing environment that includes discrimination and violence. There is a need for evidence-based MSM HIV prevention interventions that address HIV risk in the context of these psychosocial issues. This study consists of formative qualitative work followed by the development and testing of a pilot behavioral HIV prevention intervention for MSM in Chennai, India. Study goals are to maximize intervention feasibility and acceptability, estimate an effect size for a power analysis, and prepare for a full-scale trial to follow.

PHASE 1-Intervention Development. This phase involved the collection of formative data through MSM focus groups and key informant interviews to develop a subsequent pilot behavioral intervention.

PHASE 2-Open Pilot. Following Phase 1, the team conducted an open-phase non-randomized pilot of the intervention. Enrollment involved a baseline assessment that included an interviewer-administered behavioral assessment and voluntary counseling and testing for HIV and the STIs, syphilis, gonorrhea and chlamydia. Eleven MSM in Chennai then completed 6 group sessions and 4 individual sessions over 3 months. A follow-up behavioral assessment was administered upon completion of all sessions, and 6 months after baseline participants were again administered the questionnaire and HIV/STI testing.

PHASE 3-Pilot Randomized Controlled Trial. The study is currently in Phase 3, and the data articulated in this registry is for Phase 3. We are now conducting a pilot randomized controlled trial (RCT) of the intervention among 6 "batches" of 8 MSM in each group (n=48). Comparison groups (n=48) will receive the same baseline assessment and voluntary HIV/STI counseling and testing as the intervention groups. Based on Phase 2 findings, the intervention groups will meet for 4 group sessions and 4 individual sessions. Those assigned to receive the comparison condition will not receive these sessions. Participants complete the assessments approximately 3 months after randomization, and again 3 months after that.

ELIGIBILITY:
Inclusion Criteria:

* Man who has had unprotected sex with another man in past 3 months
* Resident of Tamil Nadu state, India
* Identifies as Khothi or Double-decker

Exclusion Criteria:

* Does not identify as a man (i.e. Hijra/ Ali/Transgendered)
* Under age 18
* Unable to complete or understand informed consent procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Safren, PhD, Principal Investigator — Massachusetts General Hospital, Boston, Massachusetts, United States; Beena E. Thomas, PhD, Principal Investigator — Tuberculosis Research Centre, Chennai, India
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fenway Community Health, Boston, Massachusetts
- Tuberculosis Research Centre, Chennai, Tamil Nadu, India

REFERENCES:
- [Derived] O'Cleirigh C, Safren SA, Taylor SW, Goshe BM, Bedoya CA, Marquez SM, Boroughs MS, Shipherd JC. Cognitive Behavioral Therapy for Trauma and Self-Care (CBT-TSC) in Men Who have Sex with Men with a History of Childhood Sexual Abuse: A Randomized Controlled Trial. AIDS Behav. 2019 Sep;23(9):2421-2431. doi: 10.1007/s10461-019-02482-z. PMID 30993478

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV/STI Voluntary Counseling and Testing | Behavioral Intervention
Started | 48 | 48
Completed | 42 | 42
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV/STI Voluntary Counseling and Testing | Behavioral Intervention | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (8.1) | 28.4 (6.9) | 29 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Changes in HIV Risk Taking Behavior - Number of Condomless Sex Acts Per Participant
Description: We will examine sexual risk taking among the sample using self-report (interviewer administered) measures.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: number of unprotected sex acts
Arm/Group | HIV/STI Voluntary Counseling and Testing | Behavioral Intervention
Number analyzed (Participants) | 48 | 48
number of unprotected sex acts | 7.58 (1.36) | 3.69 (.73)
Statistical Analysis 1: Comparison: HIV/STI Voluntary Counseling and Testing vs Behavioral Intervention; Intent to treat analysis; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Mixed effects Poisson regression; log(Incident Risk Ratio) = -.95, 95% CI 2-sided [-1.47 to -.44]

2. Secondary Outcome: Acquisition of STIs - Number of Participants That Acquired STIs
Description: We will test for locally relevant STIs at baseline and 6 months.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | HIV/STI Voluntary Counseling and Testing | Behavioral Intervention
Number analyzed (Participants) | 48 | 48
participants | 14 | 8
Statistical Analysis 1: Comparison: HIV/STI Voluntary Counseling and Testing vs Behavioral Intervention; Intent to treat analysis; Test type: Superiority or Other; p = .239, Chi-squared; Chi-square statistic = 1.39

3. Secondary Outcome: Changes in Psychosocial Mediators
Description: We will examine the degree to which hypothesized mediators change differentially across the experimental and control arms.
Time Frame: up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | HIV/STI Voluntary Counseling and Testing | Behavioral Intervention
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No